CLINICAL TRIAL: NCT06448052
Title: The Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Transplantation in Aging-related Low-grade Inflammation Patients' Pro-inflammatory Cytokines: a Single-group, Open-label, Phase I/II Clinical Trial
Brief Title: Umbilical Cord Mesenchymal Stem Cell for Aging-related Low-grade Inflammation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nguyen Ton Ngoc Huynh (Other)
Responsible Party: Sponsor-Investigator, Nguyen Ton Ngoc Huynh, Medical doctor, DNA International Hospital
Organization: DNA International Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 133/QĐ-BYT
Record Dates: First submitted 2024-06-01; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Disease; Aging Problems; Obese; Lipid Metabolism Disorders; Diabetes
Keywords: mesenchymal stem cell; low-grade inflammation; Inflammaging; Obese; dislipidemia; diabetes
MeSH Terms: conditions — Obesity; Lipid Metabolism Disorders; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: a single-group, open-label, phase I/II clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UC-MSC transplantation (Experimental): Participants will receive two intravenous infusions of 100 million umbilical cord mesenchymal stem cells on days 0 and 90.
  Interventions: Biological: umbilical cord mesenchymal stem cell

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cell — A total of 100 million single cells were suspended in 0.9% sterile saline solution and given intravenously at a 5-ml/min rate for 45 min. All patients will get two intravenous autologous infusions on days 0 (D0) and 90 (D90).

SUMMARY:
The goal of this single-group, open-label, phase I/II clinical trial is to evaluate the safety and efficacy of the transplantation of umbilical cord mesenchymal stem cells in aging-related low-grade inflammation patients' pro-inflammatory cytokines. The main questions to answer are:

* Is the transplantation of umbilical cord mesenchymal stem cells in aging-related low-grade inflammation patients safe?
* Comparison of the expression levels of pro-inflammatory cytokines (IL-1α/β, TNF-α/β, IL-6, IL-11, IL-18, IFN-γ) in the patient's blood before (day 0), after 90 days, and after 180 days of cell transplantation.
* Comparison of the expression levels of anti-inflammatory cytokines (IL-10, TGFβ, IL-1) in the patient's blood before (day 0), after 90 days, and after 180 days of cell transplantation.
* Comparison of the inflammation balance by the ratios of pro-inflammatory cytokines to anti-inflammatory cytokines in the patient's blood before (day 0), after 90 days, and after 180 days of cell transplantation.
* Comparison of the HbA1C index in the diabetes patient's blood before (day 0), after 90 days, and after 180 days of cell transplantation.
* Comparision of the indices of Cholesterol, Triglyceride, LDLc, HDLc in the dislipidemia patient's blood before (day 0), after 90 days, and after 180 days of cell transplantation.
* Comparison of the BMI in the obese patient's blood before (day 0), after 90 days, and after 180 days of cell transplantation.
* Determination of adverse effect frequency in the patients before (day 0), during, after 90 days, and after 180 days of cell transplatation.

Participants will receive two intravenous infusions of 100 million umbilical cord mesenchymal stem cells on days 0 and 90. The patient will be monitored for safety and measured as per the study protocol until day 180.

DETAILED DESCRIPTION:
Inflamm-aging is associated with the rate of aging and is significantly related to diseases such as Alzheimer's disease, Parkinson's disease, atherosclerosis, heart disease, and age-related degenerative diseases such as type II diabetes and osteoporosis. This study aims to evaluate the safety and efficiency of Umbilical cord mesenchymal stem cell (UC-MSC) transplantation in aging-related low-grade inflammation patients. This study is a single-group, open-label, phase I clinical trial in which patients treated with 2 infusions (100 million cells i.v) of UC-MSC were evaluated in inflamm-aging patients who concurrently had highly proinflammatory cytokines and 2 of the following 3 diseases: diabetes, dyslipidemia, and obesity. The treatment effects were evaluated based on plasma cytokines related to inflammation, HbA1C index in diabetes patients, the levels of of Cholesterol, Triglyceride, LDLc, HDLc in dislipidemia patients, BMI in obese patients. The patient will be monitored for safety during the study protocol according to the Common Terminology Criteria for Adverse Events (CTCAE) V5, NIH. The assessment of the effectiveness at days 0, 90, and 180 after cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40-64 years
* TNF-α index > 11 pg/ml and IL6 index > 1.23 pg/ml
* Possesion of at least two of the following three comorbidities: diabetes, dyslipidemia, and obesity
* Stable use of medications for the previous 3 months to treat the previously mentioned comorbidities
* Agreement to participate in the study and to comply with the research examination and evaluation process

Exclusion Criteria:

* Patients with coagulopathy
* History of or current severe heart failure
* Acute respiratory disease at the time of screening
* Patients with cancer or other acute illness requiring treatment
* History of allergy to anesthetics and antibiotics
* Currently/planning to participate in another clinical trial during the study period
* Possessing additional conditions or circumstances that make it difficult to provide treatment, according to the researcher Pathology of disease in the exclusion criteria was defined according to the Guidelines of the Ministry of Health of Vietnam.

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Adverse effect | From the patients enrolled in the study until 30 days after the study ended.
  Adverse effect will be monitored according to Common Terminology Criteria for Adverse Events (CTCAE) V5, NIH.
Serve adverse effect | From the patients enrolled in the study until 30 days after the study ended.
  Serve adverse effect will be monitored according to Common Terminology Criteria for Adverse Events (CTCAE) V5, NIH.

SECONDARY OUTCOMES:
the expression levels of pro-inflammatory cytokines | Before (day 0), after 90 days, and after 180 days of cell transplantation
  Patients peripheral blood withdraws to measure the levels of IL-1α/β (pg/mL), TNF-α/β (pg/mL), IL-6 (pg/mL), IL-11 (pg/mL), IL-18 (pg/mL), IFN-γ (pg/mL) by a suitable kit test.
the expression levels of anti-inflammatory cytokines | Before (day 0), after 90 days, and after 180 days of cell transplantation
  Patients peripheral blood withdraws to measure the levels of IL-10 (pg/mL), TGFβ (pg/mL), IL-1 (pg/mL) by a suitable kit test.
the inflammation balance | Before (day 0), after 90 days, and after 180 days of cell transplantation
  Calculation of the ratios of pro-inflammatory cytokines to anti-inflammatory cytokines in patients
Effect in diabetes patient | Before (day 0), after 90 days, and after 180 days of cell transplantation
  Diabetes patients peripheral blood withdraws to measure the levels of HbA1C (%) by a suitable kit test.
Effect in dislipidemia patient | Before (day 0), after 90 days, and after 180 days of cell transplantation
  Dislipidemia patients peripheral blood withdraws to measure the levels of of Cholesterol (mg/dL), Triglyceride (mg/dL), LDLc (mg/dL), HDLc (mg/dL) by a suitable kit test.
Effect in obese patient | Before (day 0), after 90 days, and after 180 days of cell transplantation.
  Obese patients will monitor their weight and calculate their BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen TN Huynh, MD, Principal Investigator — DNA International General Hospital, Ho Chi Minh City 700000, Vietnam
Locations (1):
- DNA International Hospital, Ho Chi Minh City, District 05, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anticipate date at the end of 2026
Access Criteria: For research only